CLINICAL TRIAL: NCT05435898
Title: Comprehensive Assessment and Digital-health Based Intervention on Early-stage Cardiovascular Organ Damage and Cardiovascular Risk in Chinese: An All-comer Registry Study
Brief Title: Assessment and Digital-health Based Intervention on Subclinical Organ Damage and Cardiovascular Risk in Chinese
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, Director of Cardiac Center, Shanghai 10th People's Hospital
Other Study IDs: NSS_2
Record Dates: First submitted 2022-06-23; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Cardiovascular Diseases; Cardiovascular Morbidity; Subclinical Organ Damage; Digital Health
Keywords: Coronary Heart Disease; Arterial stiffness; Left ventricular hypertrophy; Left ventricular diastolic dysfunction; Intima-media thickness; Cardiovascular events
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Hypertrophy, Left Ventricular; Ventricular Dysfunction, Left

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum, Stool sample and Urine sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To comprehensively evaluate subclinical organ damage of Chinese adults and its association with future cardiovascular disease and events.

To observe the significance of intervention based on digital health in preventing the onset and/or progression of subclinical organ damage and cardiovascular disease and events.

DETAILED DESCRIPTION:
In this project, we will register outpatients with cardiovascular diseases and healthy subjects for cardiovascular health check-up in the cardiovascular research clinic of our hospital, comprehensively evaluate their cardiovascular risk factors, subclinical organ damage and cardiovascular diseases at baseline. For participants who is willing to go further, a digital-based intervention will be provided for them to improve their knowledge and behaviour on cardiovascular health. For all participants, their status on subclinical organ damage, cardiovascular diseases and events will be followed within five years. The primary outcome is the composite endpoints of cardiovascular adverse events including acute coronary syndrome, myocardial infarction, heart failure, cardiovascular death. The secondary outcomes include individual cardiovascular adverse events, all-cause mortality, subclinical organ damage including cardiac damage (left ventricular hypertrophy and diastolic dysfunction), renal damage (chronic kidney disease, microalbuminuria), and vascular damage (arterial stiffness, plaques, intima-median thickening, retina arteriosclerosis). By doing these, we will be able to build a registry study and to reveal the epidemiology of subclinical organ damage, validate the association between subclinical organ damage and cardiovascular events in Chinese, and explore the significance of digital-based intervention in the prevention from subclinical organ damage and cardiovascular diseases and events.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older
* willing to participate the study and sign informed consent
* available for long-term follow-up

Exclusion Criteria:

* severe heart disease (NYHA IV)
* stage 4 or 5 CKD
* malignant tumors or with life expectancy less than 5 years
* stroke within 3 months
* refuse to participate the study or not available for long-term follow up

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All healthy subjects having cardiovascular health check-up and patients with cardiovascular diseases in the cardiovascular research clinic of our hospital are eligible for this study
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
composite endpoint of cardiovascular events | 5 years
  rate of subject with myocardial infarction, stroke, heart failure, cardiovascular death

SECONDARY OUTCOMES:
Individual cardiovascular events | 5 years
  rate of subject with individual components of composite endpoint
all cause mortality | 5 years
  rate of death
New on-set subclinical organ damage | 5 years
  Rate of subject with new on-set subclinical organ damage. Subclinical organ damage evaluated contains heart (left ventricular hypertrophy and diastolic dysfunction), kidneys (chronic kidney disease, microalbuminuria), vasculature (arterial stiffness, carotid plaque, intima-media thickness), and eye background (arteriosclerotic retinopathy).

CONTACTS AND LOCATIONS:
Overall Officials: Yi Zhang, PhD, MD, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Shanghai Tenth People's Hospital, Tongji University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang B, Gao Y, Zhao Y, Jia P, Han J, Li H, Zhang Y, Xu Y. Prognostic Value of Angiography-Derived Index of Microcirculatory Resistance in Patients with Coronary Artery Disease Undergoing Rotational Atherectomy. Rev Cardiovasc Med. 2023 Apr 27;24(5):131. doi: 10.31083/j.rcm2405131. eCollection 2023 May. PMID 39076748
- [Derived] Hou J, Li M, Han J, Yu S, Jia X, Sun F, Zhang Y. Northern Shanghai Study II: systematic assessment and management of early organ damage and its role in preventing and reducing cardiovascular risk-protocol of a prospective study. BMJ Open. 2023 Dec 30;13(12):e073423. doi: 10.1136/bmjopen-2023-073423. PMID 38159946
- [Derived] Wang B, Gao Y, Zhao Y, Xu C, Zhao S, Li H, Zhang Y, Xu Y. The spectrum of angiography-derived IMR according to morphological and physiological coronary stenosis in patients with suspected myocardial ischemia. Clin Cardiol. 2023 May;46(5):502-511. doi: 10.1002/clc.23999. Epub 2023 Mar 1. PMID 36855931